CLINICAL TRIAL: NCT00237510
Title: A Pilot Study of the Efficacy and Tolerability of Terazosin for the Treatment of Antidepressant-Induced Excessive Sweating
Brief Title: Pilot Study of Terazosin in Treatment of Antidepressant Induced Excessive Sweating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05U.84
Record Dates: First submitted 2005-10-11; First posted 2005-10-12 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Antidepressant Induced Excessive Sweating
Keywords: Antidepressant induced excessive sweating
MeSH Terms: interventions — Terazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: terazosin
  Other Names: Hytrin

SUMMARY:
This study is based on the hypothesis that terazosin, a blocker of alpha-1 receptors, will be effective in reducing excessive sweating caused by antidepressant treatment, and will have minimal adverse effects.

DETAILED DESCRIPTION:
Sweating is a common and bothersome side effect of treatment with antidepressants. Most or all antidepressants have been clearly shown to cause excessive sweating. It is unclear to what extent excessive sweating caused by antidepressants becomes less or goes away with time. In many instances, it continues to be a problem even after 6 or more months on the antidepressant.

There is no generally accepted treatment for excessive sweating. This study has been designed to study whether terazosin is effective in reducing antidepressant-induced sweating, and whether it is well-tolerated and acceptable to patients. In addition, secondary objectives of this study are to determine the time taken for patients to respond to terazosin, the usual doses needed for improvement, and the extent of reduction in sweating. This information will not only help doctors in using terazosin for this purpose in their patients, but will help in designing further studies of this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a Depressive disorder (Diagnostic and Statistical Manual of Mental Disorders - IV-TR)
* Presence of excessive sweating by self-report
* The excessive sweating started after initiation of an antidepressant and, if treatment with the antidepressant was interrupted, did not persist for more than 4 weeks during that interruption
* Treatment with the antidepressant is deemed to be clinically necessary due to substantial benefit from this antidepressant, and failure to respond to or tolerate an alternative
* Excessive sweating has persisted for at least 4 weeks prior to baseline assessment
* The excessive sweating is rated by the patient as at least moderately bothersome.
* Episodes of excessive sweating occur at least twice a week for last 4 weeks

Exclusion Criteria:

* Presence of another known disease that could potentially cause excessive sweating
* Failure to respond to antiadrenergic (reducing activity of the sympathetic nervous system) treatment in the past
* Blood pressure less than 110 mm Hg systolic at the screening or baseline visits
* Orthostatic hypotension by history or on assessment at the screening or baseline visits (defined as a decrease of 10 mm Hg or greater after standing for 2 minutes).
* Current antihypertensive treatment
* History of significant cardiac disease, including coronary artery disease
* Current use of phosphodiesterase type 5 inhibitors: sildenafil (Viagra™), tadalafil (CialisTM), or vardenafil (LevitraTM)
* History of priapism (persistent and painful erection)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2005-05; Primary Completion 2006-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To study whether terazosin 1 to 5 mg/ day is effective in reducing antidepressant-induced sweating
To determine if terazosin is tolerated and acceptable to patients as a potential treatment for antidepressant-induced sweating

SECONDARY OUTCOMES:
Determine the time-course of response, the dose-response relationship, and the magnitude of effect of treatment of antidepressant-induced sweating to assist in designing a subsequent double-blind, placebo-controlled study of this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rajnish Mago, MD, Principal Investigator — Thomas Jefferson University Department of Psychiatry and Human Behavior
Locations (1):
- Thomas Jefferson University Department of Psychiatry and Human Behavior, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Mago R, Thase ME, Rovner BW. Antidepressant-induced excessive sweating: clinical features and treatment with terazosin. Ann Clin Psychiatry. 2013 Aug;25(3):186-92. Epub 2013 May 1. PMID 23638448